CLINICAL TRIAL: NCT01372553
Title: Guilford Genomic Medicine Initiative (GGMI)
Acronym: GGMI
Status: Completed | Type: Observational
Sponsor: The Moses H. Cone Memorial Hospital (Other)
Collaborators: Duke University (Other); University of North Carolina, Greensboro (Other)
Responsible Party: Sponsor
Other Study IDs: W81XWH-05-1-0383
Record Dates: First submitted 2011-06-09; First posted 2011-06-14 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer; Ovarian Cancer; Colon Cancer; Thrombophilia
Keywords: Primary care; Family History; Risk Stratification; Cancer; Thrombosis
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Colonic Neoplasms; Thrombophilia; Neoplasms; Thrombosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Total number of project participants that completed family health history tool was 1,184.. Out of the 1,184 subjects, 75 DNA saliva samples were collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Family history risk stratification: primary care patients who receive risk stratification and clinical decision support based upon the family health history they entered in to MeTree

SUMMARY:
* Genomic medicine, using genetic information to improve health outcomes, is heralded as the answer to rising medical costs by focusing on prevention and tailored care. Despite its potential, little investigation has focused on how genomic medicine can be applied in health care. To be effective, it requires new ways to learn, deliver, and communicate medical information. It will also raise new ethical questions.
* The overall goal of Guilford Genomic Medicine Initiative (GGMI) is to identify the specific challenges in "re-structuring" an existing medical system to integrate genomic medicine, and create solutions that can be used by other medical systems, such as the extensive military medical care system. To accomplish this goal, GGMI includes the development of a large-scale genomic medicine education initiative targeted at the community, providers, and patients, and a clinical systems model to implement strategies to facilitate the integration of genomic medicine into several pilot practices.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for an upcoming well or new visit within the next 3 weeks with their primary care physician (at the two implementation clinics).

Exclusion Criteria:

* Non-english speaking
* not consentable
* adopted

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study takes place in two Primary care practices. Patient's that come in for well-visits are invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1184 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Evaluate effectiveness of family history collection and decision support for increasing appropriate referrals to genetic counselors for patients at risk of hereditary cancer syndromes | 1 year
  change in appropriate referal to genetic counseling one year before using MeTree compared to one year after.
Evaluate effectiveness of family history collection and decision support for increasing appropriate screening for breast, colon, and ovarian cancer | 1 year
  Compare rate of appropriate screening for breast, colon, and ovarian cancer one year prior to using the family history decision support tool and one year after
Evaluate effectiveness of family history collection and decision support for appropriate risk-based management of thrombosis | one year
  Evaluate rate of appropriate genetic counseling and/or genetic testing one year prior to using the family history collection and decision support tool and one year after

SECONDARY OUTCOMES:
Measure patient-related outcomes associated with using the MeTree tool | Day 1
  We assess satisfaction, comfort, anxiety, and preparedness associated with using the MeTree tool via survey immediately after completing the family history collection.
Measure physician experience with the MeTree system | 3 months
  Evaluate physicians' perceptions of satisfaction, the tool's impact on work load and its effectiveness via survey and informal interviews at 3 months.
Implementation parameters for MeTree | up to 2 years
  Part of the formative evaluation of the implementation process which includes other secondary measures as well as those related to impact on the clinic such as time to use the tool, questions asked while taking the tool, and resources and support that will be needed to implement the tool in a non-study environment

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey S Ginsburg, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Cone Health, Greensboro, North Carolina, United States

REFERENCES:
- [Background] Orlando LA, Buchanan AH, Hahn SE, Christianson CA, Powell KP, Skinner CS, Chesnut B, Blach C, Due B, Ginsburg GS, Henrich VC. Development and validation of a primary care-based family health history and decision support program (MeTree). N C Med J. 2013 Jul-Aug;74(4):287-96. PMID 24044145
- [Background] Orlando LA, Hauser ER, Christianson C, Powell KP, Buchanan AH, Chesnut B, Agbaje AB, Henrich VC, Ginsburg G. Protocol for implementation of family health history collection and decision support into primary care using a computerized family health history system. BMC Health Serv Res. 2011 Oct 11;11:264. doi: 10.1186/1472-6963-11-264. PMID 21989281
- [Result] Orlando LA, Wu RR, Beadles C, Himmel T, Buchanan AH, Powell KP, Hauser ER, Henrich VC, Ginsburg GS. Implementing family health history risk stratification in primary care: impact of guideline criteria on populations and resource demand. Am J Med Genet C Semin Med Genet. 2014 Mar;166C(1):24-33. doi: 10.1002/ajmg.c.31388. Epub 2014 Mar 10. PMID 24616329
- [Result] Wu RR, Himmel TL, Buchanan AH, Powell KP, Hauser ER, Ginsburg GS, Henrich VC, Orlando LA. Quality of family history collection with use of a patient facing family history assessment tool. BMC Fam Pract. 2014 Feb 13;15:31. doi: 10.1186/1471-2296-15-31. PMID 24520818
- [Result] Beadles CA, Ryanne Wu R, Himmel T, Buchanan AH, Powell KP, Hauser E, Henrich VC, Ginsburg GS, Orlando LA. Providing patient education: impact on quantity and quality of family health history collection. Fam Cancer. 2014 Jun;13(2):325-32. doi: 10.1007/s10689-014-9701-z. PMID 24515581
- [Result] Wu RR, Orlando LA, Himmel TL, Buchanan AH, Powell KP, Hauser ER, Agbaje AB, Henrich VC, Ginsburg GS. Patient and primary care provider experience using a family health history collection, risk stratification, and clinical decision support tool: a type 2 hybrid controlled implementation-effectiveness trial. BMC Fam Pract. 2013 Aug 6;14:111. doi: 10.1186/1471-2296-14-111. PMID 23915256